CLINICAL TRIAL: NCT02589080
Title: Phantom Limb Pain: Efficacy of Non-invasive Sensory Feedback Through the Prosthesis
Acronym: EPIONE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University Hospital (Other)
Collaborators: Aalborg University Hospital (Other); University of Freiburg (Other); Université Montpellier (Other); Indiana University School of Medicine (Other); Ecole Polytechnique Fédérale de Lausanne (Other); Universitat Autonoma de Barcelona (Other); Catholic University of the Sacred Heart (Other); Aalborg University (Other)
Responsible Party: Principal Investigator, Goran Lundborg, Professor Göran Lundborg, Lund University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPIONE-LU
Record Dates: First submitted 2015-10-11; First posted 2015-10-28 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Phantom Limb Pain
MeSH Terms: conditions — Phantom Limb

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Non-invasive sensory feedback (Experimental)
  Interventions: Behavioral: Non-invasive sensory feedback

INTERVENTIONS:
Behavioral: Non-invasive sensory feedback — A non-invasive simple sensory feedback system, which provides the user of a prosthetic hand with sensory feedback on the arm stump. It is mediated by air in a closed loop system connecting silicone pads on the prosthetic hand with pads on the amputation stump. The silicone pads in a "tactile display" on the amputation stump expand when their corresponding sensor-bulb in the prosthesis is touched, evoking an experience of "real touch". Most amputees experience phantom limb sensations and/or phantom limb pain, as well as residual limb stump pain. There is often a "map" of the phantom hand on the amputation stump, where pressure on specific skin areas result in evoked sensation from specific fingers in the amputated phantom hand. This map is the target for the sensory feedback.

SUMMARY:
Amputation of a limb may result from trauma or surgical intervention. The amputation traumatically alters the body image, but often leaves sensations that refer to the missing body part. In 50-80% amputees, neuropathic pain develops, also called phantom limb pain (PLP). Both peripheral and central nervous system factors have been implicated as determinants of PLP. Also, PLP may be triggered by physical (changes in the weather) and psychological factors (emotional stress). Recent evidence suggests that PLP may be intricately related to neuroplastic changes in the cortex, and that these changes may modulated by providing sensory input to the stump or amputation zone.

A non-invasive clinical trial will test the effectiveness of non-invasive pressure sensory feedback build into a hand prosthesis to alleviate phantom limb pain.

DETAILED DESCRIPTION:
During the pre-screen phase the investigators will assess whether the patient experiences referred phantom limb sensations or pain. In the case that the patient does experience referred sensations on the stump the investigators will map the areas where the sensation occurs on the stump and utilize this for placement of the surface actuators. In the opposite case, actuators will instead be placed in a matrix structure at the residual limb.

As a first step towards applying mechanical stimulation, the sensation thresholds (the level of stimulation where the subject first reports a sensation) have to be determined. The outcome of this procedure is a minimum of stimulation amplitude that can be applied for each stimulation site.

A first choice would be to use the referred map to place actuators. However, amputees have different phantom maps and also the number of areas varies.

A therapy will be defined based on the use of sensory feedback system integrated with the amputees hand prosthesis. The subject should use the hand prosthesis, with sensory feedback, for a duration of minimum 2 h per day during a 4 week period.

Preferably, the system should be used actively in normal daily activities.

ELIGIBILITY:
Inclusion Criteria:

* Transradial amputation
* Amputation should be in a stable phase
* Other treatments for PLP tried with poor result
* PLP experienced as over 6 on a visual analogue scale

Exclusion Criteria:

* Cognitive impairment
* Pregnancy
* History of active substance abuse disorder
* Acquired brain injury with residual impairment
* Intelligence disability
* Neurologic or musculoskeletal disease or other diseases that may affect the function of nervous system
* Pacemaker
* dermatologic condition

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-01; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Change in phantom Limb pain | Baseline and after 4 week treatment
  Baseline status includes: phantom limb pain assessed using visual analogue scale.

SECONDARY OUTCOMES:
Cortical reorganization | Baseline and after 4 week treatment (2 hours/day)
  MRI: Change in cortical response during sensory stimulation is examined

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik Sebelius, PhD, Principal Investigator — Lund University
Locations (1):
- Fredrik Sebelius, Lund, Sweden